CLINICAL TRIAL: NCT01512875
Title: Gastric Cancer and Helicobacter Pylori Infection in Lima, Peru: The Role of Water Contamination
Brief Title: S1119 Peruvian H. Pylori Water Contamination Study
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: University of Michigan (Other); Hope Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: S1119
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; water contamination; Lima, Peru

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- biopsy proven H. pylori: Patient must have lived in the districts of Lima, Peru listed in the protocol.

SUMMARY:
The objective of this study is to elucidate the role of drinking water derived from the public source in Lima, Peru and transmission of H. pylori infection using genotypic techniques.

DETAILED DESCRIPTION:
The objective of this study is to detect the presence of Helicobacter Pylori in the drinking water derived from the public network by molecular and genomic techniques in districts of Lima (Brena, Chorrillos, Comas, El Agustino, La Victoria, Lince, Los Olivos, Miraflores, Puente Piedra, Rimac, San Isidro, San Juan de Lurigancho, San Martin de Porres, Villa El Salvador, and Villa Maria del Triunfo) with high and low incidence of gastric carcinoma. The secondary objective of this study is to establish correlations between the findings in water and those of the stomach of patients with symptoms of dyspepsia who live in those districts.

ELIGIBILITY:
Inclusion Criteria:

* adults between the ages of 21-70 years old who have lived for more than 10 years in the Lima districts listed in protocol,
* who have a biopsy proven diagnosis of infection by H. pylori.
* participants must be in good general condition, mentally competent and able to provide informed consent;
* must not show evidence of dehydration or jaundice;
* must be willing to complete the patient questionnaires.
* participants must not have known allergies to any of the antibiotics used in the study.

Exclusion Criteria:

* pregnancy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of the following districts of Lima, Peru: Brena, Chorrillos, Comas, El Agustino, La Victoria, Lince, Los Olivos, Miraflores, Puente Piedra, Rimac, San Isidro, San Juan de Lurigancho, San Luis, San Martin de Porres, Via El Salvador, Villa Maria del Triunfo.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Detect H. pylori in public drinking water of Lima Peru | within 1 year of receving last sample
  To detect the presence of Helicobacter Pylori (H. pylori) in the drinking water derived from the public network by molecular and genomic techniques in districts of Lima, Peru (districts detailed in protocol).

SECONDARY OUTCOMES:
Correlation of H. pylori in water and those of stomachs of patients with symptoms | Within 1 year of receiving last sample
  To establish correlations between the findings in water and those of the stomach of patients with symptoms of dyspepsia who live in those districts.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Valdivieso, M.D., Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru